CLINICAL TRIAL: NCT01107002
Title: Comparison of 5 Day Embryo Transfer With 2-3 Day Transfer in Patients Who Failed to Conceive in Two or More Day 2-3 Embryo Transfer Cycle in Royan Institute
Brief Title: Comparison of 5 Day Embryo Transfer With 2-3 Day Transfer in Patients With Previous In Vitro Fertilization Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Hamid Gourabi, Chief, Royan Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Emb-006
Record Dates: First submitted 2010-04-17; First posted 2010-04-20 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2010-04

CONDITIONS: Infertility
Keywords: infertility; Embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Day 5 embryo transfer group (Experimental): Embryo will transfer at blastocyst stage (day 5 after ovum pick up)
  Interventions: Procedure: Day 5 embryo transfer group

INTERVENTIONS:
Procedure: Day 5 embryo transfer group — Embryo will transfer at blastocyst stage (day 5 after ovum pick up)

SUMMARY:
The purpose of this study is to determine whether embryo transfer on day 3 versus day 5 shows a significant difference in implantation, clinical pregnancy, live birth, miscarriage and multiple pregnancy rates among women with at least two previous IVF failures

DETAILED DESCRIPTION:
A total of 200 infertile women with at least two previous IVF failures will enroll in this prospective randomized clinical trial study and will randomly be divided into two groups. Random permuted blocks with a block size of 4 will be used to ensure randomization and complete allocation concealment.

The study protocol will be assessed by an independent institutional review board and Royan ethics committee.

Ovarian stimulation protocol will include the use of a GnRH agonist (Superfact; Aventis Pharma Deutshlan, Frankfurt, Germany) administered in the long (down-regulation) protocol and the subsequent addition of FSH (Gonal F, Sereno, Switzerland). Embryos will be initially cultured in G1.V5 medium) Vitrolife-Sweden)TM on day 1 and 2, being transferred from this medium to G2.V5 ) Vitrolife-Sweden)TM on day 3. Embryos will be transferred on day 5, depending on the degree of expansion of the blastocyst.

Main outcome measures will be implantation, clinical pregnancy and live birth rates.

ELIGIBILITY:
Inclusion Criteria:

* Age fewer than 40
* Normal uterine cavity and patent tubes by either hysterosalpingogram or laparoscopy and hysteroscopy
* Two previous or more failed IVF/ICSI cycles

Exclusion Criteria:

* Women with submucous myoma
* Women with intra mural or subserous myoma greater than 3 cm
* Women with Endometriosis or Endometrioma
* Hydrosalpinx

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy rate | 6-8 weeks after oocyte retrieval
Live birth rate | After 37 weeks of gestational age

SECONDARY OUTCOMES:
Implantation rate | 4 weeks after embryo transfer
Miscarriage rate | 18 weeks after fertilization

CONTACTS AND LOCATIONS:
Overall Officials: Mahnaz Ashrafi,, MD, Principal Investigator — Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org